CLINICAL TRIAL: NCT03360123
Title: Oral Anxiolysis for the Older Pediatric Patient-Which Medication is Preferred?
Brief Title: Comparison of Triazolam and Midazolam for Anxiolysis During Dental Treatment in the Pediatric Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Whitney Eichholz, Pediatric Dental Resident, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRO17080173
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Dental Anxiety
MeSH Terms: interventions — Midazolam; Triazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midazolam Hydrochloride 2Mg/mL Syrup (Active Comparator): The participants in this arm will receive midazolam+nitrous oxide at the 1st dental appointment.
  Dosage: Midazolam: Midazolam HCl Syrup 0.5mg/kg (Max: 15mg) taken 10-15 minutes prior to dental treatment.
  Interventions: Drug: Midazolam Hydrochloride 2Mg/mL Syrup
- Triazolam 0.125 MG (Active Comparator): The participants in this arm will receive triazolam+nitrous oxide at the 1st dental appointment. Dosage: Triazolam: 0.125mg tablet taken 30 minutes prior to dental treatment.
  Interventions: Drug: Triazolam 0.125 MG

INTERVENTIONS:
Drug: Midazolam Hydrochloride 2Mg/mL Syrup — Midazolam HCl Syrup 0.5mg/kg (Max: 15mg) taken 10-15 minutes prior to dental treatment.
  Arms: Midazolam Hydrochloride 2Mg/mL Syrup
Drug: Triazolam 0.125 MG — Triazolam: 0.125mg tablet taken 30 minutes prior to dental treatment.
  Arms: Triazolam 0.125 MG

SUMMARY:
This study will evaluate the perceptions of the effects of two anxiolytic medications commonly used during dental treatment in patients weighing 40 kilograms or more.

DETAILED DESCRIPTION:
Midazolam and nitrous oxide are commonly used in pediatric patients requiring anxiolysis during dental treatment. Triazolam and nitrous oxide are commonly used in adult patients requiring anxiolysis during dental treatment. The participants in this study are patients already scheduled for 2 sedation appointments to complete their dental treatment. The medications are both benzodiazepines that have similar risks, neither medication has greater adverse effects than the other. This study will evaluate the perceptions of the effects of the medications via a parent survey and chart review. The goal of the study is to determine which anxiolytic medication is perceived to provide a better sedation experience for older pediatric patients based on parent perception of the medication's effects and the patient's behavior during dental treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Weigh 40 kilograms or more.
2. 2/4 or 3/4 Frankl Behavioral Rating at their evaluation appointment.
3. Dental treatment that requires two sedation appointments. Dental treatment that requires sedation includes: fillings, crowns, pulpotomies and/or extractions.
4. Between the ages of 7-17 years old.

Exclusion Criteria:

1. Patients taking any of the following medications will be excluded from the study: Atripia, cimetidine, diltiazem, erythromycin, fluconazole, grapefruit juice, isoniazid, itraconazole, ketoconazole, nefazodone, rifampicin, ritonavir, fusidic acid, idelalisisb, methadone, olanzapine, thalidomide and/or troleandomycin.
2. Pregnant patients will be excluded.
3. Patients that have HIV-1 that is being treated with a protease inhibitor will be excluded.
4. Patients with a MTHFR mutation will be excluded.
5. Patients with acute narrow angle glaucoma will be excluded.
6. Patients that have had a previous adverse, paradoxical or allergic reaction to any benzodiazepines will be excluded from the study.
7. Patients unable to swallow medication in tablet form.
8. Patients that do not speak English as their primary language.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2018-01-26 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-04-11 (Actual)

PRIMARY OUTCOMES:
Parent Survey | 10 minutes
  Parents will complete a 4 questions post-treatment survey after the 2nd dental appointment.
Behavior Assessment during dental treatment | 60-90 minutes
  A chart review to assess patient behavior during treatment & successful completion of treatment will be completed on secure Children's Hospital of Pittsburgh of UPMC computers and will identify the patient through a coding system that will provide no link to patient identifiers. Patient behavior will be assessed using the Frankl Behavioral Rating scale. The behavior assessment will occur during the pre-sedation period, dental treatment and recovery period, which in total will take approximately 60-90 minutes. Your child's level of cooperation, willingness to accept treatment and emotions will be documented. Successful completion of treatment is determined by whether or not the treatment plan for that appointment was completed.

CONTACTS AND LOCATIONS:
Overall Officials: Whitney Eichholz, DDS, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berthold CW, Schneider A, Dionne RA. Using triazolam to reduce dental anxiety. J Am Dent Assoc. 1993 Nov;124(11):58-64. doi: 10.14219/jada.archive.1993.0233. PMID 8227774
- [Background] Coldwell SE, Awamura K, Milgrom P, Depner KS, Kaufman E, Preston KL, Karl HW. Side effects of triazolam in children. Pediatr Dent. 1999 Jan-Feb;21(1):18-25. PMID 10029963
- [Background] Kaufman E, Hargreaves KM, Dionne RA. Comparison of oral triazolam and nitrous oxide with placebo and intravenous diazepam for outpatient premedication. Oral Surg Oral Med Oral Pathol. 1993 Feb;75(2):156-64. doi: 10.1016/0030-4220(93)90086-j. PMID 8426714
- [Background] Raadal M, Coldwell SE, Kaakko T, Milgrom P, Weinstein P, Perkis V, Karl HW. A randomized clinical trial of triazolam in 3- to 5-year-olds. J Dent Res. 1999 Jun;78(6):1197-203. doi: 10.1177/00220345990780060201. PMID 10371242
- [Background] Ehrich DG, Lundgren JP, Dionne RA, Nicoll BK, Hutter JW. Comparison of triazolam, diazepam, and placebo as outpatient oral premedication for endodontic patients. J Endod. 1997 Mar;23(3):181-4. doi: 10.1016/S0099-2399(97)80272-5. PMID 9594761
- [Background] Dionne RA, Yagiela JA, Cote CJ, Donaldson M, Edwards M, Greenblatt DJ, Haas D, Malviya S, Milgrom P, Moore PA, Shampaine G, Silverman M, Williams RL, Wilson S. Balancing efficacy and safety in the use of oral sedation in dental outpatients. J Am Dent Assoc. 2006 Apr;137(4):502-13. doi: 10.14219/jada.archive.2006.0223. PMID 16637480